CLINICAL TRIAL: NCT06600451
Title: A Retrospective Multicenter Clinical Data Collection to Evaluate the Safety, Performance, and Clinical Benefits of NobelProcera® Zirconia Implant Bridges from 4 to 14 Units in Daily Dental Practice
Brief Title: A Retrospective Data Collection on NobelProcera® Zirconia Implant Bridges from 4 to 14 Units.
Status: Active, not recruiting | Type: Observational
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-1690
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dental Prosthesis, Implant-Supported
Keywords: dental prosthesis; NobelProcera; implant supported prosthesis; zirconia bridge
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients treated with NobelProcera Zr Implant Bridge (4-14-unit): Patients partially and fully edentulous in need of the implant supported dental prosthesis treated with NobelProcera Zr Implant Bridge (4-14-unit) from June 2020.
  Device is CE and available on the market in May 2020.
  Interventions: Other: observational study, no intervention is required

INTERVENTIONS:
Other: observational study, no intervention is required — Retrospective chart review, investigators provides data after reviewing patient's existing medical record; no interaction with patients is required.
  Patients were treated as per standard of care

SUMMARY:
This is a retrospective multicenter data collection in which clinical and radiographic data on implant zirconia bridges are collected from partially or fully edentulous subjects consecutively treated with at least one 4- to 14-unit NobelProcera® Zirconia Implant Bridge. This data collection will be conducted in up to 11 centers (see Appendix I) and will include between 150 to 200 subjects.

The aim of this retrospective multicenter data collection is to evaluate the safety, performance, and clinical benefits of NobelProcera® Zirconia Implant Bridges (4 to 14 units) in daily dental practice.

ELIGIBILITY:
Inclusion Criteria:

* Subject was at least 18 years old at the time of treatment,
* Subjects treated with at least one NobelProcera® Zirconia Implant Bridge (4- to 14-unit supported by 2 to 10 implants).

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated with at least one NobelProcera Zirconia Implant Bridge from 4- to 14-unit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
complications | from bridge placement to last follow-up (up to 36 months follow-up)
  biological and technical complications

CONTACTS AND LOCATIONS:
Locations (1):
- Nobel Biocare Sevices AG, Kloten, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided